CLINICAL TRIAL: NCT03377101
Title: A Randomized Phase II Trial of Fulvestrant and Palbociclib in Combination With Copanlisib (FPC) Versus Fulvestrant and Palbociclib Alone (FP) for Endocrine Resistant, Hormone Receptor Positive, HER2 Negative Metastatic Breast Cancer (FPC vs FP)
Brief Title: Fulvestrant and Palbociclib With or Without Copanlisib in Treating Patients With Hormone Receptor Positive, HER2 Negative, Stage IV Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: change in study design.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-02320; NCI-2017-02320 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10194 (Other: Duke University - Duke Cancer Institute LAO); 10194 (Other: CTEP); UM1CA186704 (NIH)
Record Dates: First submitted 2017-12-18; First posted 2017-12-19 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Estrogen Receptor Positive; HER2/Neu Negative; Progesterone Receptor Positive; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: interventions — copanlisib; Fulvestrant; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (fulvestrant, palbociclib) (Active Comparator): Patients receive fulvestrant IM on days 1 and 15 of course 1 and day 1 of subsequent courses and palbociclib PO on days 1-21. Courses repeat every 28 days in absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fulvestrant; Other: Laboratory Biomarker Analysis; Drug: Palbociclib
- Arm I (fulvestrant, palbociclib, copanlisib) (Experimental): Patients receive fulvestrant IM on days 1 and 15 of course 1 and day 1 of subsequent courses, palbociclib PO on days 1-21, and copanlisib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Drug: Fulvestrant; Other: Laboratory Biomarker Analysis; Drug: Palbociclib

INTERVENTIONS:
Drug: Copanlisib — Given IV
  Other Names: BAY 80-6946; PI3K Inhibitor BAY 80-6946
  Arms: Arm I (fulvestrant, palbociclib, copanlisib)
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Palbociclib — Given PO
  Other Names: Ibrance; PD-0332991; PD-332991

SUMMARY:
This randomized phase II trial studies the side effects and how well fulvestrant and palbociclib with or without copanlisib work in treating patients with hormone receptor positive, HER2 negative, stage IV breast cancer. Fulvestrant, palbociclib, and copanlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety profile of fulvestrant + palbociclib + copanlisib (FPC) and determine the recommended phase II treatment dose (RPTD).

II. To determine if FPC is superior to fulvestrant + palbociclib (FP) using progression-free survival (PFS) as an endpoint.

SECONDARY OBJECTIVES:

I. To assess the objective response rate (ORR = partial response [PR] + complete response [CR]) and clinical benefit rate (CBR = PR + CR + stable disease [SD] >= 6 months) of FPC versus (vs.) FP.

II. To compare the median PFS between FPC and FP arms in the following subgroups: tumor PIK3CA/PTEN altered (PIK3CA mutation or PTEN mutation/PTEN loss) and tumor PIK3CA/PTEN not altered (wild type PIK3CA and PTEN and without PTEN loss).

TERTIARY OBJECTIVES:

I. To evaluate copanlisib pharmacokinetics (PK) when administered in combination with FP.

II. To assess the median PFS in the following molecularly defined subgroups treated with either FPC or FP: tumor PIK3CA mutation vs. not, tumor PTEN mutation/PTEN loss vs. not, circulating tumor (ct) deoxyribonucleic acid (DNA) PIK3CA mutation vs. not, ctDNA PI3K/PTEN mutation vs. not, and ctDNA ESR1 mutation vs. not.

III. To evaluate ctDNA mutations at baseline and over time for response predictors at baseline, and clonal evolution associated with treatment.

IV. To assess resistance mechanisms to FP and FPC at baseline and at disease progression.

V. To examine the molecular effects of FP and FPC on tumor and circulating markers.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive fulvestrant intramuscularly (IM) on days 1 and 15 of course 1 and day 1 of subsequent courses, palbociclib orally (PO) on days 1-21, and copanlisib intravenously (IV) over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in absence of disease progression or unacceptable toxicity.

ARM II: Patients receive fulvestrant IM on days 1 and 15 of course 1 and day 1 of subsequent courses and palbociclib PO on days 1-21. Courses repeat every 28 days in absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed estrogen receptor (ER) and/or progesterone receptor (PR) positive, HER2 negative or non-amplified breast cancer that is stage IV, with measurable or non-measurable disease; ER/PR positivity is defined as at least 1% positive or Allred score of at least 3
* All patients must agree to provide archival tumor material for research and must agree to undergo research tumor biopsy before treatment if presence of easily accessible lesions (judged by the treating physician); for patients with bone only disease, or patients without easily accessible lesions for the baseline research biopsy, availability of archival tumor material (2 x 4-5 micron section unstained slides, plus 15-20 x 10 micron section unstained slides or a tumor rich block) from previous breast cancer diagnosis or treatment is required for PTEN and PIK3CA analysis
* No more than 1 prior chemotherapy in the metastatic setting; there is no limit on prior lines of endocrine therapy; (for patients enrolling to the safety run-in portion of the study, prior fulvestrant, CDK4/6 inhibitor, and everolimus is allowed)
* For patients enrolling to the randomized phase II portion of this study, demonstrated resistance to prior endocrine therapy in the metastatic setting is required; this is defined as:

  * Progressed on prior endocrine therapy in the metastatic setting or
  * Relapsed on adjuvant endocrine therapy or
  * Relapsed within 12 months of completing adjuvant endocrine therapy or
  * If received adjuvant CDK4/6 inhibitor, relapsed at least 2 years after completion of adjuvant CDK4/6 inhibitor
* Washout from prior systemic anti-cancer therapy of at least 3 weeks or 5 half-lives of the drug before the start of study treatment; washout from prior radiation therapy of at least 2 weeks before the start of the study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL collected no more than 7 days before starting study treatment
* Platelets >= 75,000/mcL collected no more than 7 days before starting study treatment
* Hemoglobin >= 8.0 g/dL collected no more than 7 days before starting study treatment
* Total bilirubin =< 1.5 x institutional upper limit of normal (=< 3 x institutional upper limit of normal for patients with Gilbert syndrome) collected no more than 7 days before starting study treatment
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (=< 5 x institutional upper limit of normal for patients with liver involvement) collected no more than 7 days before starting study treatment
* Glomerular filtration rate >= 40 mL/min/1.73 m^2 according to the Modification of Diet in Renal Disease (MDRD) abbreviated formula collected no more than 7 days before starting study treatment
* Lipase =< 1.5 x ULN collected no more than 7 days before starting study treatment
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x ULN collected no more than 7 days before starting study treatment
* Glycosylated hemoglobin (HbA1c) =< 8.5% collected no more than 7 days before starting study treatment
* Left ventricular ejection fraction (LVEF) >= 50%
* Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that their medication dose and INR/PTT is stable
* Prophylactic antiemetics may be administered according to standard practice; the routine use of standard antiemetics, including 5-HT3 blockers, such as granisetron, ondansetron, or an equivalent agent, is allowed as needed
* Patients may be postmenopausal or premenopausal women
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after the last dose of copanlisib; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of copanlisib administration
* For patients enrolling to the safety run-in portion of the study, a history of treated brain metastases is allowed if there is no disease progression symptomatically and by imaging within 28 days prior to registration and if the patient is off steroids
* Ability to understand and willing to sign a written informed consent document

Exclusion Criteria:

* For patients enrolling to the randomized phase II portion of the study, prior treatment with a CDK4/6 inhibitor or fulvestrant, or a PI3K inhibitor in the metastatic setting is not allowed
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1 with the exception of alopecia)
* Immunosuppressive therapy is not allowed while on study
* Patients who are receiving any other investigational agents
* Receiving anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Patients with brain metastasis are not eligible for the randomized phase II portion of the study; for the safety run-in portion of the study, patients with progressive brain metastases should be excluded; for patients enrolling to the randomized phase II portion of the study, patients with a history of brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to copanlisib, PI3K inhibitors, or other agents used in study
* The concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's wort) are not permitted from 14 days prior to enrollment until the end of the study; other medications that are prohibited while on copanlisib treatment:

  * Herbal medications/preparations (except for vitamins)
  * Anti-arrhythmic therapy other than beta blockers or digoxin
* Systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not permitted while on study; previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days prior to the computed tomography (CT)/magnetic resonance imaging (MRI) screening; if a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose before the screening; patients may be using topical or inhaled corticosteroids; short-term (up to 7 days) systemic corticosteroids above 15 mg prednisolone or equivalent will be allowed for the management of acute conditions (e.g., treatment non-infectious pneumonitis); the use of corticosteroids as antiemetics prior to copanlisib administration will not be allowed
* Major surgical procedure or significant traumatic injury (as judged by the investigator) within 28 days before start of treatment, or have not recovered from major side effects, open biopsy within 7 days before start of treatment
* Uncontrolled intercurrent illness, including but not limited to, symptomatic congestive heart failure (> New York Heart Association [NYHA] class 2), unstable angina pectoris, new-onset angina, cardiac arrhythmia, uncontrolled hypertension despite optimal medical management, seizure disorder requiring medication, or psychiatric illness/social situations that would limit compliance with study requirements
* Proteinuria >= grade 3 as assessed by a 24 hour [h] protein quantification or estimated by urine protein: creatinine ratio > 3.5 on a random urine sample
* Myocardial infarction < 6 months before start of treatment
* History of bleeding diathesis; any hemorrhage or bleeding event >= grade 3 within 4 weeks prior to the start of study medication
* History or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function
* History of having received an allogeneic bone marrow or organ transplant
* Patients with non-healing wound, ulcer, or bone fracture
* Patients with active, clinically serious infections > grade 2 (Common Terminology Criteria for Adverse Events [CTCAE] version [v]4.0)
* Patients with uncontrolled type I or II diabetes mellitus; uncontrolled diabetes is defined as HbA1c > 8.5%
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
* Concurrent diagnosis of pheochromocytoma
* Has undergone blood or platelet transfusion < 7 days prior to start of treatment
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with copanlisib; these potential risks may also apply to other agents used in this study
* Hepatitis B (HBV) or hepatitis C (HCV); all patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus lab panel; patients positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) will be eligible if they are negative for HBV DNA, these patients should receive prophylactic antiviral therapy; patients positive for anti-HCV antibody will be eligible if they are negative for HCV ribonucleic acid (RNA)
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Cytomegalovirus (CMV) polymerase chain reaction (PCR) positive at baseline
* Patients with history of, or current autoimmune disease are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity based on the incidence, intensity, and duration of adverse events that are related to the drug combinations and occur according to according to National Cancer Institute Common Terminology Criteria for Adverse Event version 4.0 | Up to 28 days
  Adverse events will be summarized by counts and percentages, overall as well as by does levels and by patient characteristics.
Progression free survival (PFS) | From the time on study to the time of disease progression or death or end of study, whichever earlier, assessed up to 5 years
  PFS probability will be estimated by the Kaplan-Meier (KM) product limit method and survival difference will be compared between the two arms by stratified log rank test. Hazard ratio (HR) with 95% confidence interval (CI) will be estimated between the two arms from the stratified Cox proportional hazard model, without and with adjustment for patient characteristics.

SECONDARY OUTCOMES:
Objective response rate defined as proportion of response-evaluable patients who achieve complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 | Up to 5 years
  Will be estimated with a 95% exact CI and difference between the two arms will be compared by Fisher's exact test. Raw and adjusted odds ratio (OR) will be derived with 95% CI from logistic regression without and with adjustment for patient characteristics.
Clinical benefit rate defined as proportion of response-evaluable patients who achieve CR or PR or stable of disease (SD) according to RECIST v1.1 | Up to 5 years
  Will be estimated with a 95% exact CI and difference between the two arms will be compared by Fisher's exact test. Raw and adjusted OR will be derived with 95% CI from logistic regression without and with adjustment for patient characteristics.
Overall survival (OS) according to RECIST v1.1 | From time on study to time of death or latest follow-up, whichever earlier, assessed up to 5 years
  OS probability will be estimated by the KM product limit method and survival difference will be compared between the two arms by stratified log rank test. HR with 95% CI will be estimated between the two arms from the stratified Cox proportional hazard model, without and with adjustment for patient characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ma, Principal Investigator — Duke University - Duke Cancer Institute LAO